Brief Cognitive Behavioral Conjoint Therapy for PTSD With Adjunctive Intranasal Oxytocin (CBCT+OT)

NCT05207436

2/15/23

## **Data Analytic Plan**

Primary analyses with the intent-to-treat sample evaluated change in PTSD symptoms and relationship satisfaction using weekly session, baseline, and post-treatment data analyzed with multilevel linear growth models in the *R* package lme4 and a Kenward-Roger small samples correction. To account for dyadic interdependence, time was nested within individuals and individuals were nested within couples. Analyses included two-intercept models, which produce separate slope and intercept estimates for PTSD+ veterans and non-PTSD+ partners, and a separate interaction model to test for differences between slope and intercept estimates for veterans and partners. PTSD data was composed of veteran PCL-5 and partner/collateral PCL-5 scores. Relationship satisfaction data were CSI-4 scores for both partners; at baseline and post-treatment, the four items comprising the CSI-4 were extracted from the CSI-32 to be included in growth curve analyses.